CLINICAL TRIAL: NCT06860945
Title: Development of a Predictive Model for Sexually Transmitted Infections in Individuals Using Pre-Exposure Prophylaxis for HIV in Spain
Acronym: STI_PrEPare
Status: Recruiting | Type: Observational
Sponsor: Hospital Universitario de Valme (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Anais Corma-Gomez, Medical Doctor, PhD, Hospital Clínico Universitario de Valencia
Other Study IDs: STI_PrEP24
Record Dates: First submitted 2025-02-18; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Sexually Transmitted Infections (STIs); HIV; PrEP
Keywords: STI; HIV; PrEP; modelling; machine learning; adherence; persistence
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- STI_PrEPare: All individuals with documented initiation of daily oral PrEP, who have collected the medication at least once and have taken at least one pill, will be included in the study.
  The approved criteria for the use of oral PrEP in Spain, as recommended by the Spanish Gesida guidelines (GeSIDA. Recomendaciones sobre la Profilaxis Pre-Exposición para la Prevención de la Infección por VIH en España. Marzo 2023. Disponible en http://.gesida-seimc.org/category/guias-clinicas/otras-guias-vigentes/), are as follows:
  * People without HIV infection at the time of cohort inclusion
  * Age ≥ 16 yr who meet the following criteria:
    * MSM and transgender women with at least two of the following criteria during the last year: > 10 sexual partners; Condomless anal sex; Chemsex; PEP; ≥ 1 STI
    * Sex worker women who report non-habitual use of condoms.
    * Cisgender males/females, who report condomless and present at least two of the same criteria as MSM and transgender.
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No Intervention: Observational Cohort

SUMMARY:
Objective: To develop and validate a predictive model for acquiring sexually transmitted infections (STIs) in individuals using HIV pre-exposure prophylaxis (PrEP) within the national program providing this strategy.

Methods: Ambispective cohort study, multicentric (23 Spanish hospitals). All PrEP users, with follow-up within the program, will be included. Entry into the program will be considered as the baseline visit. From there, patients are followed quarterly, following the national protocols for monitoring PrEP users in Spain. At each visit, diagnosis of different STIs (serum, pharyngeal swab, urethral or urine sample, rectal swab, endocervical/vaginal swab, ulcer) is performed. Primary outcome variable: development of an STI (Yes/No). The following STIs will be considered: syphilis, Neisseria gonorrhoeae (NG) infection, Chlamydia trachomatis (CT) infection, lymphogranuloma venereum (LGV), Mycoplasma genitalium (MG) infection, genital herpes, hepatitis A, hepatitis B, hepatitis C, HIV infection, and MPOX. Secondary outcome variable: number of diagnosed STIs. In order to determine factors associated with acquiring an STI, multivariate analyses will be conducted using logistic regression. The best models will be analyzed in the validation population. To compare the models, we will follow the Bayesian approach suggested by Benavoli et al.

ELIGIBILITY:
Inclusion Criteria:

* All individuals with documented initiation of oral PrEP (daily or event-driven regimens), who have collected the medication at least once and have taken at least one pill, will be included in the study.

The approved criteria for the use of oral PrEP in Spain, as recommended by the Spanish Gesida guidelines (GeSIDA. Recomendaciones sobre la Profilaxis Pre-Exposición para la Prevención de la Infección por VIH en España. Marzo 2023. Available at http://.gesida-seimc.org/category/guias-clinicas/otras-guias-vigentes/), are as follows:

* People without HIV infection at the time of cohort inclusion
* Age ≥ 16 yr who meet the following criteria:
* MSM and transgender women with at least two of the following criteria during the last year: > 10 sexual partners; Condomless anal sex; Chemsex; PEP; ≥ 1 STI
* Sex worker women who report non-habitual use of condoms.
* Cisgender males/females, who report condomless and present at least two of the same criteria as MSM and transgender.
* PWID with unsafe injection practices

Exclusion Criteria: none

-

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All individuals who meet the criteria for PrEP use in Spain, are over 16 years old, and have taken at least one pill.
Sampling Method: Non-Probability Sample
Enrollment: 9000 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
STI predictive model | through study completion, an average of 5 years
  Predictive model for the acquisition of sexually transmitted infections in individuals using PrEP within the national provision program for this strategy

SECONDARY OUTCOMES:
STI incidence | through study completion, an average of 5 years
  Incidence of sexually transmitted infections (STIs) in the cohort globally and by type of infection.
STI dynamics | through study completion, an average of 5 years
  Evolution of STI diagnoses during follow-up among PrEP users included in the study, both globally and by specific pathogen
asymptomatic STIs | through study completion, an average of 5 years
  Proportion of asymptomatic STIs diagnosed within the screening program.
behavioral changes | through study completion, an average of 5 years
  Sexual risk behaviors of individuals in the cohort, before and after initiating PrEP
DOXYPEP | through study completion, an average of 5 years
  Proportion of Individuals who might benefit from the 'Doxy-PEP' strategy (doxycycline use as post-exposure prophylaxis for chlamydia and syphilis)
PrEP discontinuation | through study completion, an average of 5 years
  Prevalence of oral PrEP discontinuation within a nationwide PrEP users' cohort.
Predictor of PrEP discontinuation | through study completion, an average of 5 years
  Predictors of oral PrEP discontinuation within a nationwide PrEP users' cohort.
PrEP adherence | through study completion, an average of 5 years
  Self-reported oral PrEP adherence.
Time to discontinuation | through study completion, an average of 5 years
  Time elapsed between oral PrEP initiation and oral PrEP discontinuation.
HIV incident infection | through study completion, an average of 5 years
  Incidence of HIV seroconversions
HIV incident infection | through study completion, an average of 5 years
  Profiles of those who acquire HIV while taking oral PrEP.

CONTACTS AND LOCATIONS:
Overall Officials: Anaïs Corma-Gómez, MD, PhD, Principal Investigator — Hospital Clínico Universitario de Valencia
Locations (26):
- Spain (26):
  - Hospital Universitario de Torrecárdenas, Almería
  - Hospital Universitario Puerto Real, Cadiz
  - Hospital Universitario Santa Lucía, Cartagena
  - hospital Universitario reina Sofía, Córdoba
  - Hospital Virgen de la Luz, Cuenca
  - Hospital Universitario de Elche, Elche
  - Hospital Clínico Universitario San Cecilio, Granada
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario Juan Ramón Jiménez, Huelva
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital de Jerez de la Frontera, Jerez de la Frontera
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat
  - Hospital Universitario Dr. Negrín, Las Palmas de Gran Canaria
  - Centro Sanitario Sandoval, Madrid
  - Hospital Fundación Jiménez Díaz, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario La Princesa, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen de la Macarena, Seville
  - Hospital Universitario Virgen de Valme, Seville
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario de Valladolid, Valladolid
  - Hospital Universitario Álvaro Cunqueiro, Vigo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jongen VW, Zimmermann HML, Goedhart M, Bogaards JA, Davidovich U, Coyer L, de Vries HJC, Prins M, Hoornenborg E, Schim van der Loeff MF; Amsterdam PrEP Project team in the HIV Transmission Elimination Amsterdam (H-TEAM) Initiative. Can we screen less frequently for STI among PrEP users? Assessing the effect of biannual STI screening on timing of diagnosis and transmission risk in the AMPrEP Study. Sex Transm Infect. 2023 May;99(3):149-155. doi: 10.1136/sextrans-2022-055439. Epub 2022 May 18. PMID 35584898
- [Background] Tang EC, Vittinghoff E, Philip SS, Doblecki-Lewis S, Bacon O, Chege W, Coleman ME, Elion R, Buchbinder S, Kolber MA, Liu AY, Cohen SE. Quarterly screening optimizes detection of sexually transmitted infections when prescribing HIV preexposure prophylaxis. AIDS. 2020 Jul 1;34(8):1181-1186. doi: 10.1097/QAD.0000000000002522. PMID 32205724
- [Background] van Wifferen F, Hoornenborg E, Schim van der Loeff MF, Heijne J, van Hoek AJ. Cost-effectiveness of two screening strategies for Chlamydia trachomatis and Neisseria gonorrhoeae as part of the PrEP programme in the Netherlands: a modelling study. Sex Transm Infect. 2021 Dec;97(8):607-612. doi: 10.1136/sextrans-2020-054741. Epub 2021 Jan 11. PMID 33431605
- [Background] McManus H, Grulich AE, Amin J, Selvey C, Vickers T, Bavinton B, Zablotska I, Vaccher S, Jin F, Holden J, Price K, Yeung B, Cabrera Quichua G, Ogilvie E, McNulty A, Smith D, Guy R. Comparison of Trends in Rates of Sexually Transmitted Infections Before vs After Initiation of HIV Preexposure Prophylaxis Among Men Who Have Sex With Men. JAMA Netw Open. 2020 Dec 1;3(12):e2030806. doi: 10.1001/jamanetworkopen.2020.30806. PMID 33355675
- [Background] Traeger MW, Schroeder SE, Wright EJ, Hellard ME, Cornelisse VJ, Doyle JS, Stoove MA. Effects of Pre-exposure Prophylaxis for the Prevention of Human Immunodeficiency Virus Infection on Sexual Risk Behavior in Men Who Have Sex With Men: A Systematic Review and Meta-analysis. Clin Infect Dis. 2018 Aug 16;67(5):676-686. doi: 10.1093/cid/ciy182. PMID 29509889
- [Background] Ayerdi O, Orviz E, Valls Carbo A, Fernandez Pineiro N, Vera Garcia M, Puerta Lopez T, Ballesteros Martin J, Rodriguez Martin C, Baza Caraciolo B, Lejarraga Canas C, Perez-Garcia JA, Carrio D, Garcia Lotero M, Ferreras Forcada M, Gonzalez Polo M, Raposo Utrilla M, Delgado-Iribarren A, Del Romero-Guerrero J, Estrada Perez V. Incidence of sexually transmitted infections and screening models among pre-exposure prophylaxis users. Enferm Infecc Microbiol Clin (Engl Ed). 2024 Dec;42(10):570-576. doi: 10.1016/j.eimce.2024.03.004. Epub 2024 Mar 16. PMID 38492988
- [Background] Traeger MW, Guy R, Asselin J, Patel P, Carter A, Wright EJ, Grulich A, McManus H, Fairley CK, Chow EPF, McNulty A, Finlayson R, Bell C, Owen L, Marshall L, Russell D, O'Donnell D, Donovan B, Hellard ME, Stoove MA; Australian Collaboration for Coordinated Enhanced Sentinel Surveillance of Sexually Transmissible Infections and Blood Borne Viruses (ACCESS) Study Group. Real-world trends in incidence of bacterial sexually transmissible infections among gay and bisexual men using HIV pre-exposure prophylaxis (PrEP) in Australia following nationwide PrEP implementation: an analysis of sentinel surveillance data. Lancet Infect Dis. 2022 Aug;22(8):1231-1241. doi: 10.1016/S1473-3099(22)00175-X. Epub 2022 May 25. PMID 35643090
- [Background] Traeger MW, Cornelisse VJ, Asselin J, Price B, Roth NJ, Willcox J, Tee BK, Fairley CK, Chang CC, Armishaw J, Vujovic O, Penn M, Cundill P, Forgan-Smith G, Gall J, Pickett C, Lal L, Mak A, Spelman TD, Nguyen L, Murphy DA, Ryan KE, El-Hayek C, West M, Ruth S, Batrouney C, Lockwood JT, Hoy JF, Hellard ME, Stoove MA, Wright EJ; PrEPX Study Team. Association of HIV Preexposure Prophylaxis With Incidence of Sexually Transmitted Infections Among Individuals at High Risk of HIV Infection. JAMA. 2019 Apr 9;321(14):1380-1390. doi: 10.1001/jama.2019.2947. PMID 30964528
- [Background] Hoornenborg E, Coyer L, Achterbergh RCA, Matser A, Schim van der Loeff MF, Boyd A, van Duijnhoven YTHP, Bruisten S, Oostvogel P, Davidovich U, Hogewoning A, Prins M, de Vries HJC; Amsterdam PrEP Project team in the HIV Transmission Elimination AMsterdam (H-TEAM) Initiative. Sexual behaviour and incidence of HIV and sexually transmitted infections among men who have sex with men using daily and event-driven pre-exposure prophylaxis in AMPrEP: 2 year results from a demonstration study. Lancet HIV. 2019 Jul;6(7):e447-e455. doi: 10.1016/S2352-3018(19)30136-5. Epub 2019 Jun 6. PMID 31178284
- [Background] Drak D, Mcmanus H, Vickers T, Heron JE, Vaccher S, Zablotska I, Guy R, Bavinton B, Jin F, Grulich AE, Bloch M, O'Connor CC, Gracey DM; Expanded PrEP Implementation in Communities New South Wales (EPIC-NSW) research group. Renal impairment in a large-scale HIV preexposure prophylaxis implementation cohort. AIDS. 2021 Nov 15;35(14):2319-2326. doi: 10.1097/QAD.0000000000003035. PMID 34310371
- [Background] Baeten JM, Donnell D, Ndase P, Mugo NR, Campbell JD, Wangisi J, Tappero JW, Bukusi EA, Cohen CR, Katabira E, Ronald A, Tumwesigye E, Were E, Fife KH, Kiarie J, Farquhar C, John-Stewart G, Kakia A, Odoyo J, Mucunguzi A, Nakku-Joloba E, Twesigye R, Ngure K, Apaka C, Tamooh H, Gabona F, Mujugira A, Panteleeff D, Thomas KK, Kidoguchi L, Krows M, Revall J, Morrison S, Haugen H, Emmanuel-Ogier M, Ondrejcek L, Coombs RW, Frenkel L, Hendrix C, Bumpus NN, Bangsberg D, Haberer JE, Stevens WS, Lingappa JR, Celum C; Partners PrEP Study Team. Antiretroviral prophylaxis for HIV prevention in heterosexual men and women. N Engl J Med. 2012 Aug 2;367(5):399-410. doi: 10.1056/NEJMoa1108524. Epub 2012 Jul 11. PMID 22784037
- [Background] Grant RM, Anderson PL, McMahan V, Liu A, Amico KR, Mehrotra M, Hosek S, Mosquera C, Casapia M, Montoya O, Buchbinder S, Veloso VG, Mayer K, Chariyalertsak S, Bekker LG, Kallas EG, Schechter M, Guanira J, Bushman L, Burns DN, Rooney JF, Glidden DV; iPrEx study team. Uptake of pre-exposure prophylaxis, sexual practices, and HIV incidence in men and transgender women who have sex with men: a cohort study. Lancet Infect Dis. 2014 Sep;14(9):820-9. doi: 10.1016/S1473-3099(14)70847-3. Epub 2014 Jul 22. PMID 25065857
- [Background] Grant RM, Lama JR, Anderson PL, McMahan V, Liu AY, Vargas L, Goicochea P, Casapia M, Guanira-Carranza JV, Ramirez-Cardich ME, Montoya-Herrera O, Fernandez T, Veloso VG, Buchbinder SP, Chariyalertsak S, Schechter M, Bekker LG, Mayer KH, Kallas EG, Amico KR, Mulligan K, Bushman LR, Hance RJ, Ganoza C, Defechereux P, Postle B, Wang F, McConnell JJ, Zheng JH, Lee J, Rooney JF, Jaffe HS, Martinez AI, Burns DN, Glidden DV; iPrEx Study Team. Preexposure chemoprophylaxis for HIV prevention in men who have sex with men. N Engl J Med. 2010 Dec 30;363(27):2587-99. doi: 10.1056/NEJMoa1011205. Epub 2010 Nov 23. PMID 21091279

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-02-11): https://cdn.clinicaltrials.gov/large-docs/45/NCT06860945/Prot_SAP_000.pdf
  • Informed Consent Form (2024-09-16): https://cdn.clinicaltrials.gov/large-docs/45/NCT06860945/ICF_001.pdf